CLINICAL TRIAL: NCT02091635
Title: Efficacy of Motilitone on Gastric Accommodation in Healthy Adult Patients: Evaluation Using MRI Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Poong-Lyul Rhee, Clinical Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Motilitone
Record Dates: First submitted 2014-03-06; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Dyspepsia
Keywords: accommodation, emptying, motilitone
MeSH Terms: conditions — Dyspepsia | interventions — Sugars; Tablets; DA-9701

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motilitone (Active Comparator): Eligible subjects were randomly allocated in a 1 : 1 ratio to receive either 60 mg motilitone (motilitone group) or placebo (placebo group) three times daily (before meals) for 5 days (days 1-5).
  Interventions: Drug: Placebo (for Motilitone)
- Placebo (for Motilitone) (Placebo Comparator): Eligible subjects were randomly allocated in a 1 : 1 ratio to receive either 60 mg motilitone (motilitone group) or placebo (placebo group) three times daily (before meals) for 5 days (days 1-5).
  Interventions: Drug: Motilitone

INTERVENTIONS:
Drug: Placebo (for Motilitone) — Eligible subjects were randomly allocated in a 1 : 1 ratio to receive either 60 mg motilitone (motilitone group) or placebo (placebo group) three times daily (before meals) for 5 days (days 1-5).
  Other Names: Sugar pill manufactured to mimic Motilitone 60mg tablet
  Arms: Motilitone
Drug: Motilitone — Eligible subjects were randomly allocated in a 1 : 1 ratio to receive either 60 mg motilitone (motilitone group) or placebo (placebo group) three times daily (before meals) for 5 days (days 1-5).
  Other Names: DA-9701
  Arms: Placebo (for Motilitone)

SUMMARY:
Functional dyspepsia (FD) is a disorder characterized by chronic or recurrent upper abdominal pain or discomfort in the absence of a specific structural cause. Improving gastric accommodation and prokinetic effect seem to be an attractive physiological target in patients with FD. Motilitone (Dong-A ST, Yongin, Korea) is a new herbal drug that was launched in December 2011 in Korea for treating patients with FD. The current study aims to evaluate effects of motilitone on gastric accommodation and emptying after a meal in a group of healthy volunteers using three-dimensional gastric volume measurements by magnetic resonance imaging (MRI). Healthy volunteers are randomly allocated to receive either motilitone or placebo in a double blinded manner. After 5 days of treatment, subjects undergo gastric MRI. The primary endpoint is gastric accommodation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 20 and 70 years of age without upper abdominal pain or discomfort and a structural abnormality on upper gastrointestinal (GI) endoscopy performed within the preceding 6 months were eligible for the trial.

Exclusion Criteria:

* Patients were excluded if they met any of the following criteria:

  1. any functional GI disease or previous abdominal surgery
  2. diabetes mellitus under insulin or oral anti-hyperglycemic agent treatment
  3. significant cardiopulmonary diseases or any malignancies
  4. significant renal (serum creatinine level ≥ 1.5 × the upper normal limit) or liver disease (serum aspartate aminotransferase and alanine aminotransferase levels ≥ 2.5 × the upper normal limits
  5. taking medications that may alter gastric function within 2 weeks prior to the start of the study
  6. pregnancy or lactation
  7. females with inadequate contraception during the study period
  8. contraindications to MRI (e.g., cardiac pacemaker or metallic aneurysm clip)
  9. allergic history to motilitone
  10. other conditions likely to interfere with study procedures, as judged by the investigator

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in total gastric volume (TGV) after the test meal | This outcome is measured on day 7 after 5days of treatment. The change is defined as difference between TGV 15min after the test meal and at the pre-test meal.

SECONDARY OUTCOMES:
Gastric emptying (GE) rate | This outcome is measured on day 7 after 5 days of treatment
Change in proximal TGV after the test meal | This outcome is mesured on day 7 after 5 days of treatment. The change is defined as difference between proximal TGV 15 min after the test meal and at the pre-test meal.
Change in proximal to distal TGV ratio after the test meal | This outcome is measured on day 7 after 5 days of treatment. The change is defined as difference between proximal to distal TGV ratio 15 min after the test meal and at the pre-test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Min YW, Min BH, Kim S, Choi D, Rhee PL. Effect of DA-9701 on Gastric Motor Function Assessed by Magnetic Resonance Imaging in Healthy Volunteers: A Randomized, Double-Blind, Placebo-Controlled Trial. PLoS One. 2015 Sep 24;10(9):e0138927. doi: 10.1371/journal.pone.0138927. eCollection 2015. PMID 26402448